CLINICAL TRIAL: NCT02544971
Title: Neurofeedback Therapeutic Intervention For Post-Traumatic Stress Disorder Patients Compared To Treatment As Usual
Acronym: NFTIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0215-15-TLV
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NF-N group (Experimental): Neurofeedback in a neutral context
  Interventions: Behavioral: Neurofeedback
- NF-T group (Active Comparator): Neurofeedback in a trauma-related context
  Interventions: Behavioral: Neurofeedback
- Control group (Active Comparator): Treatment as usual
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Neurofeedback — Neurofeedback is based on the learned change in a particular neural signal or a combination of neural signals when feedback and reward of these signals are repeatedly presented to the organism. Thus, individuals learn to modulate their neural activity through a closed NF loop.
  Arms: NF-N group; NF-T group
Other: Control — Treatment as usual
  Arms: Control group

SUMMARY:
Post-traumatic stress disorder (PTSD) is a common debilitating disorder that affects many individuals exposed to aversive events. The severity of PTSD symptoms is positively correlated with amygdala activation. More severe PTSD symptoms following exposure to stressful events, are associated with amygdala hyper-responsivity prior to exposure. A possible intervention for PTSD is Neurofeedback (NF) - a treatment method based on learned self-modulation of neural activity in response to feedback of neural signal. Previous work in our lab established a NF training procedure that utilizes the temporal abilities of EEG with the spatial advantages of fMRI. Further work based on this method using the amygdala BOLD signal (EEG-finger-print, EFP) has demonstrated a potential for improving the ability to self-regulate amygdala activity and to improve emotional regulation in a healthy population. The current study aims to investigate the potential of this method as a therapeutic intervention for PTSD.

DETAILED DESCRIPTION:
Pre-treatment phase (one week) Day 1 Participants will arrive at Tel Aviv Sourasky Medical Center (TASMC) and receive an explanation regarding the study and protocol and will sign informed consent. They will then be asked to fill demographic and psychological questionnaires assessing emotion regulation abilities (ERQ), state and trait anxiety (STAI), and questionnaires measuring symptoms of stress, anxiety and depression such as BDI. They will also be interviewed using clinically structured interviews (SCID, CAPS).

All participants will undergo psychiatric evaluation in the trauma clinic at TASMC. The evaluation would also entail medication monitoring.

The participants would be randomized to the three groups NF-T group (N=20), NF-N group (N=20) and treatment as usual (N=20), based on: age (under/over 40) and time since traumatic event (over or under 5 years).

Day 2 All participants will undergo a brain-imaging scan to characterize brain network responses associated with emotional arousal and regulation. Participants will be scanned for functional and structural MRI, which will include ROI localizer for the neurofeedback (NF), resting state and diffusion tensor imaging (DTI). Following which participants of the NF treatment groups will have 1 session of real-time-functional MRI-electric fingerprint neurofeedback (rt-fMRI-EFP NF) session.

Prior to this session a research staff member will explain the course of the MRI testing to the participant, and will enter with the participants into the mock simulator to verify that he or she is lying on their back properly and feel comfortable. During scanning the patient will be presented with visual and auditory stimuli, as well as short video clips. Auditory presentation: stimuli will be heard via MRI -compatible headphones. Visual displays: the participants will view the stimuli through a mirror and projected onto a screen in the magnet room. In between blocks the participants will be given time to rest. Participants will be asked to avoid moving as much as possible during the scans.

The total duration of testing, from participant arrival to departure, will take approximately 90-180 minutes (20-30 minutes to fill out forms and undergo training, 30 minutes for explanations and a break, and 60 minutes of imaging). Participants will remain in the MRI for about 60 minutes, and under no circumstances will remain longer than 90 minutes.

Treatment phase (12 weeks) The duration of the treatment phase will be 12 weeks. All groups will receive 1/2 sessions per week.

Treatment as usual sessions: Participants will obtain their regular treatment regimen (pharmacological and/or psychological) and meet with a psychologist/psychiatrist following the common practice in the clinic.

NF-EFP sessions: For the duration of each NF-EFP session the participant will be seated comfortably in front of a computer screen. A staff member will explain the goal of the meeting to the participant, present the equipment to be used and describe the course of the meeting. Following the above explanations, the staff member will place the EEG cap on the participants head and ensure that he/she feels comfortable. The EEG-NF practice will consist of about five-minute segments repeated for up to 30 minutes. During each practice segment the participant will be asked to modify visual or auditory media that provides feedback on the degree of successful brain training. For example, during visual feedback the participants will be asked to slow the speed of a skateboard presented on the computer screen or alternatively, via auditory feedback, to reduce the intensity of auditory stimuli audible through the headphones. The duration of one session is approximately 45 minutes.

NF-EFP sessions for the NF-N group: The participants will receive about one or two sessions per week as described above. All training sessions will be held in a neutral, non trauma-related, context.

NF-EFP sessions for the NF-T group: The use of trauma-related context in this group will be done gradually to ensure participants gain control over the feedback training. In the first phase that will include about 6 out of 12 sessions, the participants will train in NF sessions identical to those of the NF-N group. Participants who succeed in lowering EFP signal during training (compared to baseline) in 4 out of 6 sessions, or in the last 3 out of 5 sessions, will qualify to continue to the next phase of training. In the second phase, participants who succeed as described above, will train in the context of their traumatic story. In the first session, the participants will listen to a recording of their trauma, accompanied by one of the team members with relevant training, and will immediately train on emotional regulation using NF in a neutral context. Participants that succeed in down regulation of their EFP signal in at least one session will continue to the next trauma-context sessions. In these sessions, the feedback indicating the EFP signal would be the volume of the trauma-recording. That is, a successful reduction of EFP signal would reduce the volume of the trauma recording. Participants who don't succeed in down regulating their EFP signal (with the neutral context) immediately after listening to the trauma-recording will try again in the following NF-N session.

Midpoint assessment (one week) All participants will receive a second psychological evaluation (plus medication monitoring), will complete the questionnaires described in the pre treatment phase.

Post treatment phase (one week) Day 1 All participants will undergo a final psychiatric evaluation, and medication monitoring.

Day 2 All participants will be scanned for functional and structural MRI which will include the resting state DTI and the NF session. They will then complete the same questionnaires as in the pre treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic Post traumatic stress disorder (PTSD) (at least one year and two months since diagnosis; diagnosis according to DSM-V, or DSM-VI)
* Patients must meet the criteria for medical MRI testing set by Tel Aviv Sourasky Medical Center

Exclusion Criteria:

* Patients diagnosed with another major psychiatric disorder other than PTSD (such as schizophrenia).
* Patients diagnosed with substance abuse.
* Any aggravation of PTSD symptoms that requires hospitalization.
* Patients who are unable to commit to the duration and plan of the study.
* Patients who meet the criteria for exclusion in medical MRI scans, according to procedures set forth at MRI Medical Center in Tel-Aviv Sourasky. For example, metal that cannot be removed, orthodontal accessories connected to one's teeth, or current systemic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Decreased PTSD symptoms measured by change in psychiatric evaluation and PCL score | 1-14 weeks
  Psychiatric evaluation is based on amount and severity of symptoms according to DSM-IV/V. We will also base change in symptoms on a statistically significant change in PCL (PTSD Check List) score
Reduced amygdala reactivity measured by percent change in BOLD signal | 1-14 weeks

SECONDARY OUTCOMES:
Change in Emotion Regulation Questionnaire (ERQ) | 1-14 weeks
  36-item measure of cognitive coping strategies
Change in State/Trait Anxiety Inventory (STAI) | 1-14 weeks
  20-item measure of state & trait anxiety
Change in Beck Depression Inventory (BDI-II) | 1-14 weeks
  21-item measure of clinical depression

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, MD, PhD, Principal Investigator — Tel Aviv University Sourasky Medical Center
Locations (1):
- Whol Institute for Advanced Imaging, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel